CLINICAL TRIAL: NCT06687395
Title: Skill Retention of Advanced Airway Techniques After Simulation Training - a Randomized Prospective Study
Brief Title: Skill Retention of Advanced Airway Techniques After Simulation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Caroline Holaubek, MD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EK Nr: 1518/2024
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Educational Problems; Critical Incident; Emergencies; Airway Complication of Anesthesia
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Group 1: training model 1 - re-assessment model 1 Group 2: training model 2 - re-assessment model 1
Who Masked: Outcomes Assessor
Masking Description: pseudonymized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medium/high fidelity model (Other): Group 1: training model 1 - re-assessment model 1
  Interventions: Other: Skill training on different models
- self-made model (Other): Group 2: training model 2 - re-assessment model 1
  Interventions: Other: Skill training on different models

INTERVENTIONS:
Other: Skill training on different models — Skill training on different models (medium/high fidelity vs. self-made model)

SUMMARY:
Background: FONA (front of neck access) is a surgical airway management technique used in emergency situations, primarily as the "last option" when less invasive airway management methods have failed. The need for FONA is extremely rare, which makes regular training in this skill all the more important.

Study Objective: The objective of this study is to test "skill retention" three to four months after training on different cricothyrotomy models. The goal is to demonstrate that there is no intolerable difference in skill retention, regardless of whether FONA training is conducted on a commercially available cricothyrotomy model or on a self-made model.

Population: The study population consists of 42 participants who are randomly assigned to two groups.

Study Design: All participants begin with the same theoretical input. Following this, they complete training on their assigned practice model before undergoing an initial evaluation. Three to four months after the first evaluation, a reevaluation takes place, this time without any prior training.

Parameters: The primary outcome parameter of the study is the score achieved on the checklist. Secondary outcome parameters include the time from the start of the procedure to the first successful ventilation and subjective assessment using a Likert scale questionnaire. Possible associations between checklist results and factors such as year of training, prior experience, clinical experience, and individual items on the subjective assessment questionnaire will be presented graphically in an exploratory manner and quantified using appropriate correlation coefficients.

Hypothesis: The study aims to show that there is no intolerable difference in skill retention, regardless of whether FONA training takes place on a commercially available cricothyrotomy model or on a self-made model. This would open up the possibility of using cost-effective and readily accessible practice models for effective skill training.

DETAILED DESCRIPTION:
The study is a prospective, randomized assessment of the skill retention following a FONA (front of neck access) training. A randomized allocation is conducted, dividing participants into two groups of 21 resident physicians each from the Medical University of Vienna, Department of Anaesthesia, Intensive Care Medicine and Pain Medicine. The two groups train on two different practice models: a commercially available cricothyrotomy model (SimMan 3G, Laerdal Medical) and a self-made model based on instructions by Varaday et al. The skill retention reevaluation after three to four months takes place for all participants on the SimMan 3G.

The study begins in both groups with an identical theoretical introduction and training of FONA. Following this, all participants are given the same practice time on the model assigned to their group, before undergoing an initial evaluation. Three to four months after the initial training session and evaluation, a reevaluation is conducted in which both groups perform FONA on the SimMan 3G. The reevaluation analysis serves as the primary goal of the study, aimed at investigating the non-inferiority of the self-made model. The SimMan 3G by Laerdal was selected as it is a widely used practice model and has been described in previous studies with medium to high fidelity.

The evaluation is conducted in the form of a checklist (Difficult Airway Society), which provides a point system allowing conclusions about skill retention. Additionally, the time taken from the start to the first successful ventilation is documented and analyzed in the study as a secondary measure. After each evaluation, participants complete a questionnaire in the form of a Likert scale to assess subjective factors.

ELIGIBILITY:
Inclusion Criteria:

* Resident physicians at the Medical University of Vienna (Department of Anaesthesia, Intensive Care Medicine and Pain Medicine)
* Presence of written consent

Exclusion Criteria:

* Prior clinical experience in 'front of neck access' with more than five performed cricothyrotomies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of the training on the self-made model in terms of achieved checklist points | 3-4 months
  checklist points (0-19)

SECONDARY OUTCOMES:
years of resideny and prior experience | 3-4 months
  1) years of residency (years) / 2) prior experience with front of neck access in skill trainings (number) / 3) number of performed front of neck accesses in clinical practice (number)
time from the start of the procedure to the first successful ventilation | 3-4 months
  measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Rössler, Prof.,MD,MIH, Study Director — Department of Anaesthesia, Intensive Care Medicine and Pain Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Due to an ongoing Master thesis the dataset is not available at the moment

REFERENCES:
- [Derived] Stochlinski C, Maleczek M, Korn L, Gleiss A, Breckwoldt J, Roessler B. Skill retention of advanced airway techniques after simulation training - a randomized prospective study. BMC Med Educ. 2026 Jan 28. doi: 10.1186/s12909-026-08646-5. Online ahead of print. PMID 41606573